CLINICAL TRIAL: NCT01927406
Title: The Secondary Beneficial Effects of Prostaglandin Analog Treatment in Thyroid Eye Disease Patients.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding source unavailable
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andrea L Kossler, M.D., Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 26654
Record Dates: First submitted 2013-08-16; First posted 2013-08-22 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Thyroid Eye Disease; Ocular Hypertension; Glaucoma
Keywords: Thyroid Eye Disease; Graves' Disease; Prostaglandin Analogues
MeSH Terms: conditions — Graves Ophthalmopathy; Ocular Hypertension; Glaucoma; Graves Disease | interventions — Prostaglandins, Synthetic; Bimatoprost; Travoprost; tafluprost; Latanoprost; Timolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prostaglandin Analog vs Timolol (Experimental): In this group, with thyroid eye disease and increased intraocular pressure in both eyes, prostaglandin analog eyedrop (bimatoprost 0.01%, travoprost z 0.004%, tafluprost 0.0015% or latanoprost 0.005%) will be administered once a day, topically, into one - randomised eye. Timolol 0.5% eye drop will be administered topically in second, control eye, two times a day.
  Interventions: Drug: Prostaglandin Analog; Drug: Timolol
- Prostaglandin Analog (Experimental): In this group, with thyroid eye disease and increased intraocular pressure in only one eye Prostaglandin Analog eyedrop (bimatoprost 0.01%, travoprost z 0.004%, tafluprost 0.0015% or latanoprost 0.005%) will be administered once a day, topically, into one, affected eye.
  Interventions: Drug: Prostaglandin Analog

INTERVENTIONS:
Drug: Prostaglandin Analog — The first choice drug from group of Prostaglandin Analogues will be bimatoprost, if patient will suffer from any side effect of this drug another drug from this group will be administer. If patient turned out to cannot tolerate the prostaglandin analog therapy then the exclusion criteria will be met.
  Other Names: Bimatoprost; Travoprost Z; Tafluprost; Latanoprost
Drug: Timolol — Timolol topical eye drop will be administered in Prostaglandin Analog vs Timolol arm only, in patients with elevated intraocular pressure in both eyes.
  Other Names: Timolol maleate 0.5%
  Arms: Prostaglandin Analog vs Timolol

SUMMARY:
The purpose of this study is to evaluate the potential secondary beneficial effect of prostaglandin analogues (PA) treatment in thyroid eye disease (TED) patients. This study aims to determine if PA would change the course of the orbitopathy in TED patients by altering the progression of the common features of TED, including fatty hypertrophy, proptosis, eyelid retraction and optic nerve compression. The eyes with thyroid eye disease and elevated intraocular pressure will be randomised to the PA treatment and the other eye will serve as a control eye and will be treated with Timolol.

ELIGIBILITY:
Inclusion Criteria:

* mild or moderate to severe thyroid eye disease in one or both eyes
* age > 18 years
* informed consent
* intraocular pressure > 21 mmHg or glaucoma suspect or glaucoma diagnosed in one or both eyes
* not on current prostaglandin analog intraocular pressure lowering therapy

Exclusion Criteria:

* sight threatening thyroid eye disease
* children < 18 years old
* patients that are not compliant with treatment or follow-up
* patients already on prostaglandin analog treatment
* patients that undergo cosmetic periocular procedures during the study will be excluded from further follow up
* patients that cannot tolerate prostaglandin analog treatment.
* patients with bilateral thyroid eye disease and elevated intraocular pressures that cannot tolerate treatment with timolol or an alternative intraocular pressure lowering medication such as trusopt, combigan, cosopt.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06 (Estimated); Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in appearance of facial periorbital region at 6 months. | Baseline and 6 months

SECONDARY OUTCOMES:
Change from baseline in Hertel exophthalmometry at 3, 6, 9 and 12 months. | Baseline and 3, 6, 9 and 12 months
Change from baseline in intraocular pressure at 3, 6, 9 and 12 months. | Baseline and 3, 6, 9 and 12 months
Change from baseline in appearance of facial periorbital region at 3, 6, 9 and 12 months. | Baseline and 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L. Kossler, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States